CLINICAL TRIAL: NCT07173751
Title: A Phase III, Multisite, Randomized, Double-Blind Trial of BNT327 in Combination With Chemotherapy Versus Placebo With Chemotherapy in Patients With Previously Untreated Locally Recurrent Inoperable or Metastatic TNBC Determined Ineligible for PD(L)1 Therapy Based on PD-L1 Negative Disease
Brief Title: ROSETTA Breast-01: The Effects and Safety of Pumitamig in Patients With Triple-Negative Breast Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: BioNTech SE (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BNT327-05; 2025-521884-12-00 (EU CTIS Number)
Record Dates: First submitted 2025-09-08; First posted 2025-09-15 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Breast Neoplasms
Keywords: Metastatic TNBC; Bispecific antibody; Programmed death-ligand 1 (PD-L1); Immunotherapy; Immunotherapy in combination with chemotherapy; Combination with other investigational agents
MeSH Terms: conditions — Breast Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Gemcitabine; Carboplatin; eribulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: Pumitamig + Treatment of Physician's Choice (TPC) Chemotherapy (Experimental): Participants will be administered with pumitamig (BNT327) plus chemotherapy regimen.
  Interventions: Drug: Pumitamig; Drug: Nab-paclitaxel/Paclitaxel; Drug: Gemcitabine; Drug: Carboplatin; Drug: Eribulin
- Arm 2: Placebo + TPC Chemotherapy (Placebo Comparator): Participants will be administered with matching placebo plus chemotherapy regimen.
  Interventions: Drug: Nab-paclitaxel/Paclitaxel; Drug: Gemcitabine; Drug: Carboplatin; Drug: Eribulin; Drug: Matching placebo

INTERVENTIONS:
Drug: Pumitamig — Solution for intravenous (IV) infusion
  Other Names: BNT327; PM8002; BMS-986545
  Arms: Arm 1: Pumitamig + Treatment of Physician's Choice (TPC) Chemotherapy
Drug: Nab-paclitaxel/Paclitaxel — IV infusion
Drug: Gemcitabine — IV infusion
Drug: Carboplatin — IV infusion
Drug: Eribulin — IV infusion
Drug: Matching placebo — IV infusion
  Arms: Arm 2: Placebo + TPC Chemotherapy

SUMMARY:
This is a Phase III trial where participants will be randomized to two treatment groups, which means participants will be assigned by equal chance to a treatment group. This trial will be double-blinded, which means neither the participants nor the trial doctors will know which of the two treatments the participants actually receive. Participants will receive either the trial drug with chemotherapy or placebo (which looks like the trial drug but does not have any drug in it) with chemotherapy.

DETAILED DESCRIPTION:
The study consists of a:

1. Screening period (up to 28 days);
2. Treatment period, during which participants will receive pumitamig or placebo in combination with chemotherapy (until disease progression, the occurrence of intolerable toxicity, withdrawal, death, or trial termination [whichever comes first]);
3. Safety follow-up (FU) period (for up to 90 days after administration of the last dose of trial treatment) and survival follow-up (until the participant dies, withdraws consent for survival status follow-up, loss of contact, or sponsor decision, whichever occurs first).

Participants will be randomized 1:1 to receive either pumitamig in combination with the treatment of physician's choice (TPC) chemotherapy (Arm 1) or placebo in combination with TPC chemotherapy (Arm 2). Chemotherapy will be administered per standard of care. The randomization will be stratified based on the following factors:

* Prior treatment with cancer immunotherapy (yes versus no)
* On-trial chemotherapy regimen (paclitaxel/nab-paclitaxel versus gemcitabine plus carboplatin versus eribulin)
* Geography (East Asia versus the rest of the world [ROW])
* PD-L1 status (combined positive score [CPS] less than [<] 1 versus 1 less than or equal to [<=] CPS <10).

ELIGIBILITY:
Inclusion Criteria:

* Are considered ineligible for combination treatment with a monospecific PD(L)1 targeting immunotherapy plus chemotherapy as per their tumor PD-L1 expression status.
* Have confirmed locally recurrent inoperable or metastatic TNBC, or estrogen receptor (ER)-low, human epidermal growth factor receptor 2 (HER2)-negative breast cancer (ER and/or progesterone receptor [PgR]) 1% to 10%, HER2 immunohistochemistry [IHC] 0, 1+, or 2+ with fluorescence in situ hybridization [FISH] negative for HER2 gene amplification) documented prior to trial screening as part of standard of care.
* Have at least one measurable lesion as the targeted lesion based on RECIST v1.1.
* Have provided a tissue sample, archival or fresh, during the screening period (bone biopsies, fine needle aspiration biopsies, and samples from pleural or peritoneal fluid are not acceptable; participants with only one target lesion are not eligible to participate in the trial).
* Eastern cooperative oncology group (ECOG) performance status of 0 or 1.

Exclusion Criteria:

* Have received any of the following therapies or drugs prior to the initiation of trial:

  * Have received prior systemic anticancer therapy for advanced disease.
  * Have received prior treatment with a PD(L)-1/vascular endothelial growth factor (VEGF) bispecific antibody.
  * Have received systemic corticosteroids (at a dosage greater than 10 milligrams [mg]/day of prednisone or an equivalent dose of other corticosteroids) within 7 days prior to the initiation of trial treatment. Exception: excluding local, intranasal, intraocular, intra-articular or inhaled corticosteroids, short-term use (<= 7 days) of corticosteroids for prophylaxis (for example, prevention of contrast agent allergy) or treatment of non-autoimmune conditions (for example, delayed hypersensitivity reactions caused by exposure to allergens).
  * Have been vaccinated with live attenuated vaccine(s) within 4 weeks prior to initiation of trial treatment.
  * Have received broad-spectrum intravenous antibiotics therapy within 2 weeks prior to initiation of trial treatment.
* Are pregnant or breastfeeding or are planning pregnancy or planning to father children during the trial or within 6 months after the last dose of pumitamig or placebo.
* Have undergone major organ surgery, significant trauma, or invasive dental procedures (such as dental implants) within 28 days prior to the initiation of trial treatment or plan to undergo elective surgery during the trial. Placement of vascular infusion devices is allowed.
* Have received allogeneic hematopoietic stem cell transplantation or organ transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 558 (Estimated)
Dates: Start 2025-10-30 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) as Assessed by Blinded Independent Central Review (BICR) | Up to approximately 32 months
  PFS is defined as the time from randomization to first documented tumor progression (progressive disease assessed by BICR per response evaluation criteria in solid tumors [RECIST] v1.1), or death from any cause, whichever occurs first.
Overall Survival (OS) | Up to approximately 49 months
  OS is defined as the time from randomization to death from any cause.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) as Assessed by BICR | Up to approximately 49 months
  ORR is defined as the percentage of participants in whom a confirmed complete response (CR) or confirmed partial response (PR) as per RECIST v1.1 is assessed by BICR as best overall response.
PFS | Up to approximately 32 months
  PFS is defined as the time from randomization to first documented tumor progression (progressive disease assessed by investigator per RECIST v1.1), or death from any cause, whichever occurs first.
ORR | Up to approximately 49 months
  ORR is defined as the percentage of participants in whom a confirmed CR or confirmed PR (per RECIST v1.1) is observed as best overall response.
Duration of Response (DOR) | Up to approximately 49 months
  DOR is defined as the time from first objective response (CR or PR per RECIST v1.1) to first occurrence of objective tumor progression (progressive disease per RECIST v1.1), or death from any cause, whichever occurs first.
Disease Control Rate (DCR) | Up to approximately 32 months
  DCR is defined as the percentage of participants in whom a confirmed CR or confirmed PR or stable disease (SD) (per RECIST v1.1, SD assessed at least 6 weeks after randomization) is observed as best overall response.
PFS Rate as Assessed by BICR | At 6, 12, 18, and 24 months
PFS Rate as Assessed by Investigator | At 6, 12, 18, and 24 months
OS Rate | At 6, 12, 18, and 24 months
Occurrence of Treatment-Emergent Adverse Events (TEAEs) Including Grade Greater than or Equal to (>=) 3, Serious, and Fatal TEAEs by Relationship | From the first dose of study treatment to the 90-days after last dose of study treatment (up to approximately 57 months)
  TEAEs graded according to United Stated (US) National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0)
Occurrence of Dose Interruption, Reduction, and Discontinuation of Trial Treatment due to TEAEs (including related TEAEs) | From the first dose of study treatment to the 90-days after last dose of study treatment (up to approximately 57 months)
Change from Baseline in European Organization for Research and Treatment of Cancer (EORTC) Quality-of-Life Core 30 Questionnaire (QLQ-C30) Global Health Status/Quality-of-Life score (Items 29 and 30) | Baseline up to approximately 49 months
  Global health status or quality of life (QoL) scale ranges in score from 0 to 100 with a high scale score representing a higher response level (for example, high score for global health status/QoL is high QoL: high score for symptom scale/item is high symptomatology or problems).
Change from Baseline in EORTC QLQ-C30 Physical Functioning | Baseline up to approximately 49 months
  Physical functioning scale ranges in score from 0 to 100 with a high scale score representing a higher response level (for example, high score for functional scale is high/healthy level of functioning).
Change from Baseline in Arm Symptoms Scale of EORTC QLQ-Breast Cancer (BR)42 | Baseline up to approximately 49 months
  Arm symptom scale ranges in score from 0 to 100 with a high scale score representing a higher level of symptoms or problems.
Change from Baseline in Breast Symptoms Scale of EORTC QLQ-BR42 | Baseline up to approximately 49 months
  Breast symptom scale ranges in score from 0 to 100 with a high scale score representing a higher level of symptoms or problems.
Change from Baseline in Functional Assessment of Cancer Therapy-General Version (FACT-G) Overall Bother Item (FACT-GP5) | Baseline up to approximately 49 months
  The single-item GP5, that is "I am bothered by side effects of treatment," is rated on a 5-point Likert scale (where 1=not at all and 5=very much) by the participants. A high scale score represents worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: BioNTech Responsible Person, Study Director — BioNTech SE
Locations (8):
- United States (8):
  - Highlands Oncology Group, Springdale, Arkansas
  - Cancer Care Specialists of Illinois, O'Fallon, Illinois
  - New England Cancer Specialists, Westbrook, Maine
  - Lahey Hospital & Medical Center, Burlington, Massachusetts
  - Profound Research LLC at Michigan Hematology and Oncology Consultants, Royal Oak, Michigan
  - The West Clinic, P.C. dba West Cancer Center, Germantown, Tennessee
  - Oncology Consultants PA, Houston, Texas
  - Northwest Medical Specialties, PLLC, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No